CLINICAL TRIAL: NCT03417258
Title: Bioavailability of Phytoestrogens and Prevalence of Adenomatous Polyps in Human Colon
Brief Title: Phytoestrogens and Colonic Adenomatous Polyps
Acronym: FITOPOL
Status: Completed | Type: Observational
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, Michele Barone, Researcher, University of Bari
Other Study IDs: Policlinic Hospital, Bari
Record Dates: First submitted 2018-01-18; First posted 2018-01-31 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Intestinal Polyps
Keywords: phytoestrogens; isoflavones; adenomatous polyps; microbiome
MeSH Terms: conditions — Intestinal Polyps; Adenomatous Polyps

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Urine, feces
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with polyps: urinary phytoestrogen excretion and intestinal microbiota evaluation
- Patients without polyps: urinary phytoestrogen excretion and intestinal microbiota evaluation

SUMMARY:
INTRODUCTION: The data obtained by experimental studies about the influence of phytoestrogens on colorectal cancer (CRC) have been very promising. On the other hand, clinical trials have produced conflicting results. The literature suggests that some subclasses of phytoestrogens may have protective effects against CRC and colon adenomas, but most of these results come from population studies based on the dietary intake of phytoestrogens. On these premises, it is possible to hypothesize that the variability of the data reported in the literature may be due to the fact that the real absorption of phytoestrogens (by assessing their concentration in the serum or urine) and/or the ability of the single individual of producing equol was not evaluated.

PURPOSE: In the present study, the association between the phytoestrogens intake and the prevalence of colon adenomas was evaluated not only on the basis of the simply dietary intake but also on the measurement their intestinal absorption. Moreover, a specific evaluation of equol production by the intestinal flora was performed. Finally, intestinal bacteria involved in equol production were evaluated.

DETAILED DESCRIPTION:
MATERIALS AND METHODS: Patients with sporadic colon adenomas were enrolled in group I (case) and patients without sporadic colorectal adenomas matched for sex, age and BMI were enrolled in group II (control). All participants underwent the following evaluations: BMI, dietary history (for quantitative and qualitative analysis of dietary habits), quantitative analysis of phytoestrogens (by dietary questionnaires), medications (chronic assumption of aspirin at low doses), characteristics of the polyps (for a calculation the cancer risk), analysis of urinary excretion of phytoestrogens [by high pressure liquid chromatography (HPLC)] and intestinal flora [by mass spectrometry with Matrix Assisted Laser Desorption Ionization Time-of-Flight (MALDI-TOF) technology]. At the enrolment, patients will be invited to assume a standard quantitative of phytoestrogens at 8:00 a.am. and collect both a fecal sample and the urine of the following 24 hrs.

ELIGIBILITY:
Inclusion Criteria:

* subjects of both sexes aged between 50 and 75 years
* colonoscopy within 3 months from the study evaluation

Exclusion Criteria:

* age < 50 and > 75 years
* previous diagnosis of colon cancer or inflammatory bowel diseases (IBD)
* Hereditary intestinal tumors (FAP, HNPCC, ...)
* ongoing infections
* intake, in the last 4 weeks, of drugs that alter the intestinal bacterial flora
* creatinine clearance below 60 ml/min
* liver failure

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients (aged between 50 and 75 years) undergoing colonoscopy within 3 months from the study evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2019-04-24 (Actual)

PRIMARY OUTCOMES:
Phytoestrogen absorption | one day
  It will be evaluated on the basis of their 24h urine excretion

SECONDARY OUTCOMES:
Intestinal microbiota | one day
  It will be evaluated on fecal samples

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Di Leo, Study Chair — University of Bari
Locations (1):
- Policlinic Hospital, Bari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xu X, Harris KS, Wang HJ, Murphy PA, Hendrich S. Bioavailability of soybean isoflavones depends upon gut microflora in women. J Nutr. 1995 Sep;125(9):2307-15. doi: 10.1093/jn/125.9.2307. PMID 7666247
- [Background] Atkinson C, Frankenfeld CL, Lampe JW. Gut bacterial metabolism of the soy isoflavone daidzein: exploring the relevance to human health. Exp Biol Med (Maywood). 2005 Mar;230(3):155-70. doi: 10.1177/153537020523000302. PMID 15734719
- [Background] Jin H, Leng Q, Li C. Dietary flavonoid for preventing colorectal neoplasms. Cochrane Database Syst Rev. 2012 Aug 15;2012(8):CD009350. doi: 10.1002/14651858.CD009350.pub2. PMID 22895989
- [Background] Kocic B, Kitic D, Brankovic S. Dietary flavonoid intake and colorectal cancer risk: evidence from human population studies. J BUON. 2013 Jan-Mar;18(1):34-43. PMID 23613386
- [Background] Setchell KD, Brown NM, Lydeking-Olsen E. The clinical importance of the metabolite equol-a clue to the effectiveness of soy and its isoflavones. J Nutr. 2002 Dec;132(12):3577-84. doi: 10.1093/jn/132.12.3577. PMID 12468591

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-01-24): https://cdn.clinicaltrials.gov/large-docs/58/NCT03417258/Prot_SAP_ICF_003.pdf